CLINICAL TRIAL: NCT05972083
Title: The Efficacy of Serratus Posterior Superior Interfacial Plane Block on Postoperative Pain Control in Female Patients Underwent Mastectomy and Axillary Lymph Node Dissection: A Randomized, Prospective, Controlled Study
Brief Title: Serratus Posterior Superior Interfascial Plane Block for Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 33
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Breast Diseases
Keywords: Mastectomy and axillary dissection surgery; Postoperative pain management; Serratus Posterior Superior Interfascial Plane Block
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Intervention Model Description: There are two models for this study. The first group is the SPSIPB group. The second one is the control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The anesthesiologist who performs postoperative pain evaluation and the patient will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S = SPSIPB group (Active Comparator): A high-frequency linear US probe (11-12 MHz, Vivid Q) will be covered with a sterile sheath, and an 80 mm block needle (Braun 360°) will be used. The procedure will be performed with the patient in the lateral decubitus position. After the scapula is shifted slightly laterally, the US probe is placed sagittal at the upper corner of the spina scapula, and the serratus posterior superior muscle is visualized with the third rib. The in-plane technique will be used. The block needle will be advanced in the craniocaudal direction to enter between the serratus posterior superior and the third rib. The block location will be confirmed by injecting 5 ml of saline between the rib and the muscle. After the block location is confirmed, 30 ml of 0.25% concentration bupivacaine will be used.
  Interventions: Drug: Analgesia management; group S and C
- Group C = Control group (Other): The wound infiltration with 30 ml of 0.25% concentration of bupivacaine will be performed by the surgical team.
  Interventions: Drug: Analgesia management; group S and C

INTERVENTIONS:
Drug: Analgesia management; group S and C — Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. If the NRS score is ≥ 4, 0.5 mg kg-1 iv meperidine will be administered as a rescue analgesic. Postoperative patient evaluation will be performed by an anesthesiologist blinded to the procedure.

SUMMARY:
Regional techniques can be used for postoperative pain control following breast surgery. Ultrasound (US) guided serratus posterior superior block (SPSPB) is a new interfacial plane block defined by Tulgar et al in 2023. It is based on injection on the serratus posterior superior muscle at the level of the 2nd or 3rd rib. This block provides analgesia in conditions such as interscapular pain, chronic myofascial pain syndromes, scapulocostal syndrome, and shoulder pain. The SPS muscle is located at the C7-T2 level. It attaches to the lateral edges of the second and fifth ribs. It is innervated by the lower cervical and upper intercostal nerves. With the SPS block, these nerves are blocked and analgesia is provided.

DETAILED DESCRIPTION:
Mastectomy and axillary lymph node dissection are among the most frequently performed surgeries today, and pain control is an important problem affecting patient comfort in the postoperative period in these patients. Postoperative pain is an acute pain associated with the inflammatory process that occurs due to surgical trauma and gradually decreases with tissue healing. Several analgesic drugs such as opioids are used to prevent this pain, but these agents have many unwanted side effects. Successful postoperative analgesia occurs in the patient due to pain; it is a known fact that it prevents many of the effects such as not being able to breathe easily and delayed mobilization.

Regional techniques can be used for postoperative pain control following breast surgery. Ultrasound (US) guided serratus posterior superior block (SPSIPB) is a new interfacial plane block defined by Tulgar et al in 2023. It is based on injection on the serratus posterior superior muscle at the level of the 2nd or 3rd rib. This block provides analgesia in conditions such as interscapular pain, chronic myofascial pain syndromes, scapulocostal syndrome, and shoulder pain. The SPS muscle is located at the C7-T2 level. It attaches to the lateral edges of the second and fifth ribs. It is innervated by the lower cervical and upper intercostal nerves. With the SPS block, these nerves are blocked and analgesia is provided.

In the cadaveric study of Tulgar et al., it was determined that the spread of serratus posterior superior interfacial plane block; 7-10 intercostal levels on the left side only in the superficial fascia of the trapezius muscle. Spread dye was observed at intercostal levels, absent on the right. There was prominent staining on both sides of the deep trapezius muscle. Both the surface and skin of the rhomboid major were clearly stained, while the rhomboid minor was only stained in the skin. SPSP block will provide successful analgesia in procedures involving the thoracic region such as chronic myofascial pain, breast surgery, thoracic surgery, and shoulder surgery.

In this study, our aim is to investigate the efficacy of US-guided SPSIPB for postoperative analgesia management after mastectomy and axillary lymph node dissection surgery. Our primary aim is to compare postoperative pain scores (NRS), and our secondary aim is to evaluate the need for rescue analgesics, block-related complications, dermatome level, and side effects (allergic reaction, nausea, vomiting) associated with opioid use.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for mastectomy and axillary dissection surgery under general anesthesia

Exclusion Criteria:

* receiving anticoagulant treatment,
* known study drugs allergy,
* opioid addiction
* infection of the skin at the site of the block,
* pregnancy or lactation,

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients who will undergo breast surgery will be included
Enrollment: 60 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Pain scores (Numerical rating scale-NRS) | Changes from baseline pain scores at postoperative 1, 2, 4, 8, 16, and 24 hours
  The primary aim is to compare NRS at the postoperative 1st h. Postoperative pain assessment will be performed using the NRS (0 = no pain, 10 = the most severe pain felt). The NRS scores will be recorded

SECONDARY OUTCOMES:
Need for rescue analgesia (meperidine) | Postoperative 24 hours period
  The secondary aim is to compare rescue analgesia used in the postoperative 24 h.
Adverse events | Postoperative 24 hours period
  The secondary aim is to compare the adverse events (nausea, vomiting, itching) related to opioid use.
Dermatomal analyses | Postoperative 1st hour
  The secondary aim is to evaluate the dermatomal coverage of SPSIPB in Group S. The dermatomal coverage will be evaluated with a pinprick test.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Korkmaz AO, Bozkurt NN, De Cassai A, Torres AJ, Elsharkawy H, Alici HA. Serratus Posterior Superior Intercostal Plane Block: A Technical Report on the Description of a Novel Periparavertebral Block for Thoracic Pain. Cureus. 2023 Feb 3;15(2):e34582. doi: 10.7759/cureus.34582. eCollection 2023 Feb. PMID 36883093
- [Background] Ciftci B, Alver S, Ahiskalioglu A, Bilal B, Tulgar S. Serratus posterior superior intercostal plane block for breast surgery: a report of three cases, novel block and new indication. Minerva Anestesiol. 2023 Nov;89(11):1054-1056. doi: 10.23736/S0375-9393.23.17432-3. Epub 2023 Jun 1. No abstract available. PMID 37272274